CLINICAL TRIAL: NCT05004597
Title: Three-dimensional Normative Craniofacial Morphologic Development of Healthy Infants During the First Year of Life
Brief Title: 3D Craniofacial Morphologic Development of Healthy Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pangyunchou, Assistant professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201701939B0
Record Dates: First submitted 2021-07-28; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Development, Infant; IMAGE; Craniofacial Asymmetry; Plagiocephaly
Keywords: craniofacial development; growth chart
MeSH Terms: conditions — Plagiocephaly

STUDY DESIGN:
Intervention Model Description: all subjects longitudinally received 3D image
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infants longitudinally received three dimensional photo (Experimental): A series of 3D craniofacial photos were captured using a 3dMDHead System (3dMD, Atlanta, GA, USA) within 7 days before or after the age of 1, 2, 4, 6, 9, and 12 months
  Interventions: Other: three dimensional photography using a 3dMDHead System (3dMD, Atlanta, GA, USA)

INTERVENTIONS:
Other: three dimensional photography using a 3dMDHead System (3dMD, Atlanta, GA, USA) — A series of 3D craniofacial photos were captured using a 3dMDHead System (3dMD, Atlanta, GA, USA) within 7 days before or after the age of 1, 2, 4, 6, 9, and 12 months.

SUMMARY:
Healthy infants were enrolled to receive three dimensional craniofacial photography regularly at their age of one month, two month, four month, six month, nine month and twelve month. All the image data was analyzed to reveal infants' craniofacial development.

DETAILED DESCRIPTION:
Importance The development of craniofacial morphology in the first year of life is critical, especially when analyzed with longitudinal 3-dimensional photographs.

Objective To evaluate the development of the craniofacial region in healthy infants in the first year of life and provide treatment guidelines for craniofacial deformities such as orofacial clefts and deformational plagiocephaly.

Design, Setting, and Participants Three-dimensional (3D) photographs of included participants were captured using a 3dMD system. Participants were grouped by sex and age (1, 2, 4, 6, 9, and 12 months). We placed 32 craniofacial anatomical landmarks on 3D craniofacial photos. The thin-plate spline algorithm and closest-point matching were applied to transform a symmetric 3D template into a series of scanned images to calculate 3D composite heads at different ages.

Main Outcomes and Measures Average craniofacial meshes were calculated for each group. The growth patterns of the following anthropometric indices were determined: craniofacial height, depth, width, volume, body height, weight, body mass index (BMI), and head circumference.

ELIGIBILITY:
Inclusion Criteria:

* Asian ethnicity
* healthy infants
* full-term

Exclusion Criteria:

* growth curve <3%
* premature
* congenital craniofacial anomaly
* hormonal anomaly.
* chromsomal anomaly
* thyroid anomaly
* bone anomaly

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — 15 males, and 15 females
Enrollment: 30 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
craniofacial height | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
craniofacial height | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
craniofacial height | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
craniofacial height | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
craniofacial height | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
craniofacial height | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
craniofacial depth | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
craniofacial depth | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
craniofacial depth | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
craniofacial depth | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
craniofacial depth | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
craniofacial depth | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
craniofacial width | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
craniofacial width | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
craniofacial width | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
craniofacial width | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
craniofacial width | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
craniofacial width | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
craniofacial volume | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
craniofacial volume | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
craniofacial volume | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
craniofacial volume | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
craniofacial volume | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
craniofacial volume | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
body weight | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
body weight | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
body weight | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
body weight | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
body weight | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
body weight | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
body height | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
body height | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
body height | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
body height | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
body height | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
body height | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
body mass index (BMI) | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
body mass index (BMI) | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
body mass index (BMI) | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
body mass index (BMI) | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
body mass index (BMI) | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
body mass index (BMI) | at infants' age of 12 month-old
  measurement of craniofacial anthropometry
head circumference | at infants' age of 1 month-old
  measurement of craniofacial anthropometry
head circumference | at infants' age of 2 month-old
  measurement of craniofacial anthropometry
head circumference | at infants' age of 4 month-old
  measurement of craniofacial anthropometry
head circumference | at infants' age of 6 month-old
  measurement of craniofacial anthropometry
head circumference | at infants' age of 9 month-old
  measurement of craniofacial anthropometry
head circumference | at infants' age of 12 month-old
  measurement of craniofacial anthropometry

CONTACTS AND LOCATIONS:
Overall Officials: Pangyun Chou, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
three dimensional photo acquisition for newborns